CLINICAL TRIAL: NCT02002104
Title: Endothelialized ePTFE Graft by Nanobiotechnology
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201009047R
Record Dates: First submitted 2013-10-23; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: The Apparatus for Processing the Tubular Graft Modification Will be Designed and Evaluated.; The On-site Capturing of the Endothelial (Progenitor) Cells by Peptide-mediated Selective Adhesion in Vitro and in Vivo Will Also be Elucidated.; The Patency Rate of ITRI-made Artificial Blood Vessels Will be Evaluated by the Porcine Animal Model.
Keywords: Expanded polytetrafluoroethylene( ePTFE)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- EPCs: No proliferation and no differentiation on the ePTFEs
- Modified ePTFE: EPCs adherence, proliferation and differentiation on the ePTFEs.

SUMMARY:
The replacement of autologous blood vessels by artificial grafts is urgently needed in clinical applications. Expanded polytetrafluoroethylene (ePTFE) grafts are the most clinically used artificial blood vessels because of its chemical and mechanical stability. But, when used as arteriovenous (AV) grafts for haemodialysis, small diameter ePTFE grafts have a high failure rate of 40% in three years in vivo because of the functional lack of an intact endothelial cell layer. Here we developed a two-step modification including chemical etching and plasma activation to enhance the hydrophilicity of ePTFE. Peptide motifs (eg. cyclic RRE, RGD) known to bind integrins on the endothelial cells were immobilized on ePTFE grafts. Functional peptide immobilization significantly increased the adherence and growth of HUVEC cells on ePTFEs. Patch ePTFE implantation in the pig's descending aorta was used to evaluate the in vivo endothelialization of these modified ePTFE grafts. At 28 days implantation, newly formed endothelial layers on peptide-immobilized ePTFE grafts were demonstrated by SEM and histological analysis. These preliminary data showed the potential to grow an intact endothelial layer to improve the patency rate of the modified ePTFE grafts.

ELIGIBILITY:
Obtained from the peripheral blood leukocyte thick liquid (Hsinchu Blood Center, Taiwan Blood Services Fundation) Times - sampled 20 ~ 40ml / time, 2 to 3 times / month

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Native arteriovenous fistulas are not available in up to 40 percent of patients with renal dialysis. Therefore, the replacement of autologous blood vessels by artificial grafts is urgently needed. Expanded polytetrafluoroethylene( ePTFE) grafts are the most clinically used artificial blood vessels.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Isolate and expand EPCs from peripheral blood | 24 weeks
  Obtained from the peripheral blood leukocyte thick liquid (Hsinchu Blood Center, Taiwan Blood Services Fundation)

CONTACTS AND LOCATIONS:
Overall Officials: I Hui Wu, PhD, Principal Investigator — Cardiac Surgical Division, Surgical Department, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipai, Taiwan